CLINICAL TRIAL: NCT05511012
Title: Does the Therapist's Assessment of Movement Control in Low Back Pain Patients Correspond to an Objective Kinematic Modification
Acronym: LOBACOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC22.0128
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Chronic Low-back Pain
Keywords: Low back pain; Movement control; Kinematic analysis; Clinical assessment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: It is a prospective, monocentric, exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- motion control fault testing (Other): Each patient make six motion control fault tests in the same order :
  1. "waiters bow"
  2. "pelvic tilt"
  3. "one leg stance"
  4. "sitting knee extension"
  5. "rocking 4 point kneeling"
  6. "prone knee bend"
  This tests are performed three times.
  Interventions: Other: motion control fault tests

INTERVENTIONS:
Other: motion control fault tests — Patients make 6 motion control fault tests, in the same order. Each test is performed three times

SUMMARY:
* Exercise-based treatment is part of the recommendations for good practice in the treatment of low back pain (acute, sub-acute and chronic).
* The low back pain population is heterogeneous. This heterogeneity would cause the positive effects of a treatment to be canceled out by the negative effects of another part of the population.
* This polymorphism has led several authors to classify low back pain into subgroups. These subgroups constitute more homogeneous clinical pictures and would facilitate the adaptation of treatments.
* The recommendations of the American Physical Therapy Association suggest 5 subgroups of low back pain. One of them is "low back pain with movement coordination defect". In this subgroup, Luomajoki studied the reliability of different functional tests used in clinical practice. 6 out of 10 motion control fault tests show good reliability.
* The quantified analysis of the movement of low back pain patients would make it possible to determine the sensitivity of detecting an anomaly in the 6 lumbar movement control tests.

DETAILED DESCRIPTION:
* Exercise-based treatment is part of the recommendations for good practice in the treatment of low back pain (acute, sub-acute and chronic).
* The low back pain population is heterogeneous. This heterogeneity would cause the positive effects of a treatment to be canceled out by the negative effects of another part of the population.
* This polymorphism has led several authors to classify low back pain into subgroups. These subgroups constitute more homogeneous clinical pictures and would facilitate the adaptation of treatments.
* The recommendations of the American Physical Therapy Association suggest 5 subgroups of low back pain. One of them is "low back pain with movement control impairment". In this subgroup, Luomajoki studied the reliability of different functional tests used in clinical practice. 6 out of 10 motion control fault tests show good reliability.
* The quantified analysis of the movement of low back pain patients would make it possible to determine the sensitivity of detecting an anomaly in the 6 lumbar movement control tests.

LoBaCoM is a monocentric, exploratory prospective study.

The purpose is to define a kinematic (angular) threshold corresponding to an anomaly detected clinically by three therapists for each test.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years
* Common low back pain with medical prescription for rehabilitation
* Signed consent
* Be affiliated to a social security scheme
* Be able to perform the lumbar motion control failure tests

Exclusion Criteria:

* Body Mass Index greater than 30 (obesity)
* Person who does not understand French
* Pregnant woman
* Refusal to participate
* Volunteer under guardianship or curatorship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Range of compensation motion : "waiters bow" test | Day 0
  Lumbar flexion measured for test number 1 "waiters bow". Patients are filmed during the test. Videos are watched by three physiotherapists. They going to establish a diagnostic normal or abnormal
Range of compensation motion : "pelvic tilt" test | Day 0
  thoracic flexion measured for test number 2 "pelvic tilt". Patients are filmed during the test. Videos are watched by three physiotherapists. They going to establish a diagnostic normal or abnormal.
Range of compensation motion : "One leg stance" test | Day 0
  Pelvic shift measured for test number 3 "One leg stance ". Patients are filmed during the test. Videos are watched by three physiotherapists. They going to establish a diagnostic normal or abnormal.
Range of compensation motion : "sitting knee extension" test | Day 0
  Lumbar flexion measured for test number 4 "sitting knee extension". Patients are filmed during the test. Videos are watched by three physiotherapists. They going to establish a diagnostic normal or abnormal.
Range of compensation motion : "rocking 4 point kneeling" test | Day 0
  Lumbar flexion and extension measured for test number 5 "rocking 4 point kneeling ". Patients are filmed during the test. Videos are watched by three physiotherapists. They going to establish a diagnostic normal or abnormal.
Range of compensation motion : "prone knee bend" test | Day 0
  Lumbar extension measured for test number 6 "prone knee bend". Patients are filmed during the test. Videos are watched by three physiotherapists. They going to establish a diagnostic normal or abnormal

SECONDARY OUTCOMES:
Speed of execution for test 1 | Day 0
  It is measured with a camera. The camera can film one hundred pictures per second. Speed of execution is measured in seconds.
Speed of execution for test 2 | Day 0
  It is measured with a camera. The camera can film one hundred pictures per second. Speed of execution is measured in seconds.
Speed of execution for test 3 | Day 0
  It is measured with a camera. The camera can film one hundred pictures per second. Speed of execution is measured in seconds.
Speed of execution for test 4 | Day 0
  It is measured with a camera. The camera can film one hundred pictures per second. Speed of execution is measured in seconds.
Speed of execution for test 5 | Day 0
  It is measured with a camera. The camera can film one hundred pictures per second. Speed of execution is measured in seconds.
Speed of execution for test 6 | Day 0
  It is measured with a camera. The camera can film one hundred pictures per second. Speed of execution is measured in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, Finistère, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.